CLINICAL TRIAL: NCT03043950
Title: A Non-interventional Study to Assess the Safety and Efficacy of First Line Therapy With Vectibix® in Combination With FOLFIRI or FOLFOX and to Validate a Prognostic Score in Adult Patients With RAS Wild-type Metastatic Colorectal Cancer in a Real World Setting (VALIDATE)
Brief Title: Validation of a New Prognostic Score for Adult Patients With RAS Wild-type mCRC Treated With Vectibix® and FOLFIRI or FOLFOX in First Line (VALIDATE)
Acronym: VALIDATE
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-050341
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Colorectal Cancer; RAS Wild-type
Keywords: mCRC; First line; Panitumumab; mCCS Prognostic Score; Prognosis; Ras wild type
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Folfox protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low risk: Low risk according to metastatic Colorectal Cancer Prognostic Score (mCCS)
  Interventions: Drug: Panitumumab
- medium risk: Medium risk according to metastatic Colorectal Cancer Prognostic Score (mCCS)
  Interventions: Drug: Panitumumab
- high risk: High risk according to metastatic Colorectal Cancer Prognostic Score (mCCS)
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Patients will be scheduled to receive first line therapy with the combination of Panitumumab (6 mg / kg i.v, given once every two weeks) and FOLFIRI or FOLFOX, according to current SmPC.
  Other Names: + FOLFIRI or FOLFOX

SUMMARY:
A safety and efficacy study of first line therapy with Vectibix® in combination with FOLFIRI or FOLFOX to validate a prognostic score in adult patients with RAS wild-type metastatic colorectal cancer in a real world setting (VALIDATE)

DETAILED DESCRIPTION:
This is a non-interventional, prospective, open-label, single-arm, 3-cohort, multicenter study in Germany and Austria. In total, 606 patients will be enrolled in approx. 120 oncological sites (office-based medical oncologists, oncology outpatient-centers, and university hospitals) in a time period of 48 months. Of these, 202 patients with high risk, 202 patients with intermediate risk, and 202 patients with low risk, as a priori assessed by the metastatic colorectal cancer prognostic score (mCCS), will be included. Overall survival of the pre-defined prognostic groups will be analyzed as primary endpoint to validate the mCCS.

Patients have been scheduled to receive first line combination therapy with panitumumab and FOLFIRI or FOLFOX according to the current SmPC valid for Germany and Austria, respectively. Data on efficacy in terms of tumor response evaluation / survival and safety (ADRs) will be collected during first line therapy. A subset of patients participating in the 'VALIDATE-PRO' project (n=303) will be assessed for general and health-related quality of life with patient questionnaires. Biomarker status beyond RAS will be collected at baseline. The documentation of defined patient data including survival will continue until the end of the individual study participation which is latest 36 months after last patient in. The end of study will be at latest at 36 months after last patient in (LPI).

ELIGIBILITY:
Inclusion Criteria:

* Eligibility according to current SmPC
* Signed written informed consent
* Diagnosis of RAS-WT mCRC
* No prior systemic therapy in the palliative setting
* Aged 18 years or older

Exclusion Criteria:

* Any contraindication according to current SmPC
* Participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with RAS-WT mCRC scheduled for the treatment with panitumumab and FOLFIRI or FOLFOX who have not received any prior systemic antineoplastic therapy in the palliative setting.
Sampling Method: Probability Sample
Enrollment: 647 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) of pre-defined risk groups low vs. high | From date of start of first line therapy to date of death due to any cause (assessed up to 84 months)
  OS is defined as time from start of first line therapy to the date of death. For patients without date of start of first line therapy, date of informed consent will be the relevant date.

SECONDARY OUTCOMES:
Overall Survival (OS) of pre-defined risk groups low vs. intermediate | From date of start of first line therapy to date of death due to any cause (assessed up to 84 months)
  OS is defined as time from start of first line therapy to the date of death.
Overall Survival (OS) of pre-defined risk groups intermediate vs. high | From date of start of first line therapy to date of death due to any cause (assessed up to 84 months)
  OS is defined as time from start of first line therapy to the date of death.
Overall Survival (OS) | From date of start of first line therapy to date of death due to any cause (assessed up to 84 months)
  OS is defined as time from start of first line therapy to the date of death.
2-years OS Rate (2-yrs OSR) | at 24 months
  2-yrs OSR is defined as percentage of patients who are alive at 2 years after start of first line therapy.
Progression-free Survival (PFS) | From date of start of first line therapy to date of progression or death due to any cause (assessed up to 84 months)
  PFS is defined as time from start of first line therapy to first documentation of tumor progression or death due to any cause, whichever occurs first.
12-months PFS Rate (12-mos PFSR) | at 12 months
  2-yrs PFSR is defined as percentage of patients who are have not progressed or died due to any cause at 2 years after start of first line therapy.
Overall Response Rate (ORR) | From date of start of first line therapy to date of progression or death to any cause (assessed up to 84 months)
  ORR is defined as percentage of patients who achieve a partial or complete response as best response during the treatment period.
Duration of Response (DoR) | From date of start of first line therapy to date of progression or death to any cause (assessed up to 84 months)
  DoR is defined as time from first documentation of any tumor response (≥ PR) until disease progression or death due to tumor progression.
Primary and secondary resection of metastases | From date of start of first line therapy to date of death due to any cause (assessed up to 84 months)
  Data on primary and/or secondary resections of liver or lung metastases will be collected.
Antineoplastic treatment in later lines | From date of start of first line therapy to date of death due to any cause (assessed up to 84 months)
  Treatment sequences with duration will be documented.

OTHER OUTCOMES:
Patient-reported general and health-related quality of life ('VALIDATE PRO') | From date of start of first line therapy to date of progression or death due to any cause (assessed up to 84 months)
  Quality of life will be assessed with the EORTC QLQ-C30 and the EORTC Colorectal Modul QLQ-CR29 patient questionnaires during first line treatment and correlated with outcome.
Adverse Drug Reactions | From start of first line therapy until 30 days after the end of treatment with panitumumab (assessed up to 84 months)
  Adverse Drug Reactions of Panitumumab

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Marschner, Dr., Principal Investigator — Forschungs GbR Drs. Marschner, Zaiss, Kirste, Semsek
Locations (1):
- Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No